CLINICAL TRIAL: NCT00833339
Title: Novel Therapeutics in PTSD: A Randomized Clinical Trial of Mifepristone
Brief Title: Trial of Mifepristone in Combat Veterans With Posttraumatic Stress Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julia A. Golier, M.D., Clinical Director, Mental Health Patient Care Center, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 3293-08-015
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): mifepristone
  Interventions: Drug: mifepristone
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: mifepristone — 600 mg/day x 1 week
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The investigators propose to conduct a randomized double-blind, parallel-group, placebo-controlled trial of mifepristone in veterans with military-related posttraumatic stress disorder (PTSD). This study will examine the clinical, neuropsychological, and neuroendocrine effects of short-term treatment of mifepristone (600 mg/day for one week) to determine if this treatment is efficacious in improving PTSD symptoms, cognitive functioning, or other related clinical measures. Additionally, the investigators will observe whether baseline neuroendocrine activity, or other clinical or neuropsychological factors predict the response to mifepristone, and whether mifepristone-induced changes in neuroendocrine activity are associated with treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male U.S. veteran
* Subject was exposed to combat or another criterion A traumatic event during military service
* Subject meets diagnostic criteria for chronic PTSD

Exclusion Criteria:

* Veteran has a history of adrenal insufficiency or a plasma cortisol level less than 5 mcg/dl at screening
* Veteran has a moderate-severe traumatic brain injury, a history of a stroke, or another neurological illness or injury likely to impact cognitive functioning
* Veteran has diabetes mellitus, an endocrinopathy, or another major medical illness.
* Veteran is taking oral corticosteroids
* Veteran has a lifetime diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder
* Veteran is currently suicidal or otherwise is in need of urgent clinical care
* Veteran is currently receiving specialized trauma-focused psychotherapy (i.e., prolonged exposure, cognitive processing therapy or eye movement and desensitization reprocessing).
* Veteran is not willing to use effective means of birth control during the study or for 90 days after taking study medication
* Veteran has history of allergic reaction to mifepristone

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-05; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the total severity of the CAPS-2 and dichotomously defined clinical responder status. | baseline, endpoint, 4 week follow-up

SECONDARY OUTCOMES:
Change in cognitive functioning as measured by the MATRICS neuropsychological test battery and self-reported measures of depression and PTSD. | baseline, endpoint, 4 week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Golier, MD, Principal Investigator — JJP VAMC; Mount Sinai Sch of Med
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States